CLINICAL TRIAL: NCT05682599
Title: A Phase II Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Azvudine in Preventing SARS-Cov-2 Infection in Household Contacts of Individuals Infected With SARS-CoV-2 in China
Brief Title: Evaluate Azvudine in Preventing SARS-Cov-2 Infection in Household Contacts of Covid-19 in China
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Henlius Biotech (Industry)
Collaborators: Huashan Hospital (Other); Shanghai Fosun Pharmaceutical Industrial Development Co. Ltd. (Industry); Henan Genuine Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FNC-Covid201
Record Dates: First submitted 2023-01-10; First posted 2023-01-12 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — azvudine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A：Azvudine 5 mg (Experimental): Azvudine 5 mg, QD PO, D1-D7
  Interventions: Drug: Azvudine
- B：Azvudine 3 mg (Experimental): Azvudine 3 mg + placebo 2 mg, QD PO, D1-D7
  Interventions: Drug: Azvudine; Drug: Placebo
- C：placebo (Placebo Comparator): placebo 5 mg, QD PO, D1-D7
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azvudine — Azvudine is a novel nucleoside reverse transcriptase inhibitor.
  Other Names: FNC
  Arms: A：Azvudine 5 mg; B：Azvudine 3 mg
Drug: Placebo — Placebo
  Arms: B：Azvudine 3 mg; C：placebo

SUMMARY:
A Phase II Randomized, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Azvudine in Preventing SARS-Cov-2 Infection in Household Contacts of Individuals Infected with SARS-CoV-2 in China

DETAILED DESCRIPTION:
A multicentre, randomized, double-blind, placebo-controlled phase II clinical study to evaluate the efficacy and safety of Azvudine versus placebo in preventing SARS-CoV-2 infection in household contacts with SARS-CoV-2 infection individuals.Approximately 300 adults with household contact exposure to individuals with a confirmed SARS-CoV-2 infection will be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1、18-65 years old at the signing of informed consent. 2、Household contacts of individual with symptomatic COVID-19. Symptomatic COVID-19 cases (index case) to be identified as those symptomatic and recently tested (rapid antigen test or RT-PCR) positive for SARS-CoV-2 and must fulfill the following criteria 1) collection of the first positive SARS-CoV-2 test sample less than 24 hours before randomization, 2) have at least one symptom attributable to COVID-19.

3、RT-PCR test negative (with nasopharyngeal [NP] swab samples) OR rapid antigen test negative at the time of screening and without any suspicious COVID-19 symptoms within 2 weeks before randomization.

4、Subject expects to be living in the same household with the symptomatic COVID-19 cases during the whole study period.

Exclusion Criteria:

1. Subject with a history of SARS-CoV-2 vaccinations within 1 months before randomization.
2. Subject with a history of SARS-CoV-2 infection within 6 months before randomization.
3. With any serious infection requiring systemic anti-infective therapy within 14 days before randomization.
4. Allergic to the investigational agent or any components of the formulation. Pregnant or breast-feeding women.
5. Women of childbearing potential who are unwilling to practice highly effective contraception during the study, and for at least 6 months after the study; Sexually active men who are unwilling to use medically acceptable birth control during the study period.
6. Have other conditions not suitable for inclusion as judged by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-04-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Efficacy-Incidence of SARS-CoV-2 infection in 8 days | Day 2 to Day 7
  The incidence of SARS-CoV-2 infection (RT-PCR positive) up to 8 days from 2 days after administration of Azvudine for prevention of SARS-CoV-2 infection.

CONTACTS AND LOCATIONS:
Overall Officials: chen mingquan, Principal Investigator — Huashan Hospital
Locations (1):
- Huashan Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No